CLINICAL TRIAL: NCT00040326
Title: Early Randomized Surgical Epilepsy Trial
Brief Title: Early Surgical Intervention to Treat Epilepsy
Acronym: ERSET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Jerome Engel, Jr., M.D., Ph.D., UCLA School of Medicine, Department of Neurology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01NS42372
Record Dates: First submitted 2002-06-24; First posted 2002-06-25 (Estimated); Last update posted 2010-02-23 (Estimated); Status verified 2010-02

CONDITIONS: Epilepsy; Epilepsy, Temporal Lobe; Seizures
Keywords: epilepsy; mesial temporal lobe epilepsy; temporal lobe epilepsy; MTLE; seizures; anteromesial temporal resection; surgery; antiepileptic drugs; hippocampal sclerosis
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe; Seizures; Hippocampal Sclerosis | interventions — Anticonvulsants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): anteromesial temporal resection
  Interventions: Procedure: anteromesial temporal resection
- 2 (Active Comparator): antiepileptic drugs
  Interventions: Drug: antiepileptic drugs

INTERVENTIONS:
Procedure: anteromesial temporal resection — surgical treatment for epilepsy
  Arms: 1
Drug: antiepileptic drugs — pharmacotherapy
  Arms: 2

SUMMARY:
The purpose of this trial is to compare the effectiveness of early surgical intervention for mesial temporal lobe epilepsy to continued treatment with antiepileptic drugs.

DETAILED DESCRIPTION:
Mesial temporal lobe epilepsy (MTLE) is the most common form of epilepsy, and the most medically intractable. An estimated one-quarter to one-half of the 400,000 patients in the United States with intractable epilepsy have MTLE. Generally, MTLE becomes intractable in adolescence and early adulthood. Persistence of seizures during this time commonly causes adverse social and psychological consequences which can become irreversible.

The current treatment of MTLE primarily consists of medications to control seizures. Usually surgical treatment is considered only if medications are not effective. Recent studies have shown that surgery can stop disabling seizures in 60 to 70% of patients with long standing MTLE. However, to date, no research study has examined surgery performed as an early therapy.

The goal of the study is to determine if more patients treated with early surgery become seizure free and have improved quality of life compared to similar patients who continue to receive antiepileptic medication only. This study will determine the difference in seizure frequency between the two groups and the impact of the two treatments on the quality of life of the participants.

ELIGIBILITY:
Inclusion criteria:

* Intractability: Two AEDs, one of which was either Dilantin, Tegretol, Carbatrol, or Trileptal used in appropriate doses, have failed due to inefficacy, not intolerance.
* Frequency and Duration: Persistence of disabling seizures at 6 per year or greater for less than two years after onset, or after recurrence if initial treatment resulted in seizure freedom for 6 or more months.
* Age: 12 years or older at baseline visit.
* History: Simple and complex partial seizures, with or without secondarily generalized seizures beginning in childhood or later, with or without febrile convulsions earlier.
* Absence of a history of serious cerebral insult after the age of 5; a progressive neurological disorder; mental retardation (I.Q. less than 70); psychogenic seizures; focal neurological deficits other than memory disturbances; unequivocal focal extratemporal EEG slowing or interictal spikes; or lesions on neuroimaging outside of the mesial temporal area.
* Seizure semiology: Auras that occur in isolation and are not primary sensory other than olfactory or gustatory. Absence of initial focal motor movements other than automatisms or dystonic posturing. Presence of postictal confusion.
* Neurological examination: No unexplained focal or lateralized neurological deficits other than memory dysfunction.
* Baseline QOL and ancillary outcome data:
* Adolescents - QOLIE-48-AD, CHQ, CBCL, PANAS, Life Events Scale, FAC, FEICS-PC completed.
* Adults - QOLIE-82/ESI55, locus of control, PANAS, Life Events Scale, FAD, FEICS-PC completed.
* Global rating scale completed.
* Baseline ancillary outcomes completed. Psychiatric evaluation: No evidence of psychosis, current or recent substance abuse, suicidality, anorexia, or psychogenic seizures. Baseline BSI and MINI or KSADS completed.
* Neuropsychological testing: I.Q. of greater than 70. No significant focal neurocognitive dysfunction inconsistent with MRI and PET findings. Baseline neuropsychological testing completed.
* Neuroimaging: Hippocampal atrophy on MRI T1 imaging with either increased ipsilateral mesial signal on T2 imaging, or ipsilateral hypometabolism on PET (Class I), or either hippocampal atrophy on MRI only, or temporal hypometabolism on PET only (Class II).
* Absence of temporal neocortical or extratemporal lesions on MRI, or diffuse unilateral or bilateral hypometabolism on PET.
* Video-EEG Monitoring:
* If neuroimaging is Class I, ictal EEG onset is lateralized to the ipsilateral side; if neuroimaging is Class II, ictal EEG onset is focal on the ipsilateral side.
* Absence of contralateral or extratemporal ictal onset.
* Absence of persistent extratemporal, or predominant contralateral focal interictal spikes or slowing, or generalized interictal spikes.
* Absence of psychogenic seizures.
* Seizure baseline: Seizure log, seizure report forms, and seizure severity scale completed.
* IAP: In those randomized to surgery only, contralateral hemisphere can support memory.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2002-07; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be freedom from disabling epileptic seizures (complex partial and secondarily generalized seizures, and simple partial seizures that are apparent to an observer) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Engel, Jr., M.D., Ph.D., Principal Investigator — UCLA School of Medicine, Department of Neurology
Locations (12):
- United States (12):
  - Barrow Neurological Institute, Phoenix, Arizona
  - UCLA School of Medicine, Department of Neurology, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Department of Neurology, Ann Arbor, Michigan
  - University of Rochester, Department of Neurology, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Engel J Jr, McDermott MP, Wiebe S, Langfitt JT, Stern JM, Dewar S, Sperling MR, Gardiner I, Erba G, Fried I, Jacobs M, Vinters HV, Mintzer S, Kieburtz K; Early Randomized Surgical Epilepsy Trial (ERSET) Study Group. Early surgical therapy for drug-resistant temporal lobe epilepsy: a randomized trial. JAMA. 2012 Mar 7;307(9):922-30. doi: 10.1001/jama.2012.220. PMID 22396514